CLINICAL TRIAL: NCT04751890
Title: Effectiveness of a Home-based Structured Exercise Program Versus Walking Advice in Patients With Peripheral Artery Disease: a Randomized-controlled Trial
Brief Title: Structured Home-based Exercise Versus Walking Advice in Claudication Patients: a Randomized-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 898/2020/Sper/AOUFe
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Artery Disease
Keywords: exercise; rehabilitation; exercise testing
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to patients' allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured home-based exercise (Experimental): Program will include two 8-minute sessions/day (6 days/week) of intermittent walking (1-minute work and 1-minute rest while seated) at a prescribed speed converted into a walking cadence and followed at home using a metronome. The walking sessions will be preferably performed indoors at home or on a treadmill. During the study, 2 follow-up visits (at weeks 8 and 16) will be performed to evaluate patient adherence to the program and to update the exercise program with the duration of each session that remained constant. The walking intensity of each exercise regime will be progressively modified to increase the training load. The patients will be asked to fill out a daily training record indicating completion of the exercise and any associated symptoms. Patients will have the ability to contact the rehabilitation team, composed of a physician and a sports science expert, throughout the entire study period via phone.
  Interventions: Behavioral: Structured home-based exercise
- Walking advice (Active Comparator): Patients will receive advice to walk as suggested by the guidelines. In particular, a team member will recommend patients to gather almost 30 minutes of walking at least 3 times per week; when the patient will face claudication pain, he/she will be allowed to rest, and restart walking as soon as possible. A daily log to be compiled will be provided to each patients to record the amount of walk performed.
  Interventions: Behavioral: Walking advice

INTERVENTIONS:
Behavioral: Structured home-based exercise — Low-intensity interval walking program prescribed at hospital and performed at daily at home
  Arms: Structured home-based exercise
Behavioral: Walking advice — Walking advice according to the guidelines for peripheral artery disease patients
  Arms: Walking advice

SUMMARY:
A recent position paper calls for effective home-based exercise program for patients with peripheral artery disease (PAD) and claudication to be implemented in real-world care.

This randomized-controlled trial aims to test the effects on mobility, hemodynamics and cardiovascular outcomes of a structured home-based exercise program (SHB) compared to walking advice (WA) recommendation intended as usual care, in PAD patients.

Male and females PAD patients at Leriche-Fontaine's stage II and aged more than 60 years old will be enrolled. Patients will be randomized in SHB or WA groups.

Patients of SHB group will receive a prescription of a home-based walking program during serial testing sessions at the hospital. The program will include two 10-minute sessions/day (6 days/week) of intermittent walking (1-minute work and 1-minute rest while seated) at a prescribed speed converted into a walking cadence and followed at home using a metronome. Two follow-up visits (at weeks 8 and 16) will be performed to evaluate patient adherence and to update the exercise program by increasing the walking speed.

Patients randomized in WA group will receive the advice to walk as suggested by the guidelines. In particular, patients will be recommended to gather almost 30 minutes of walking at least 3 times per week; when they will face claudication pain, they will be allowed to rest and restart walking as soon as possible.

Outcome measures will be performed at the entry prior to randomization, at the end of exercise programs (6-month) and after 12-month follow up. Primary outcomes will be the pain-free walking distance and the 6-minute walking distance collected during the 6-minute walking test Secondary outcomes will include ankle-brachial index, quality of life, lower limb strength and long-term clinical outcomes including revascularization and mortality.

ELIGIBILITY:
Inclusion Criteria:

* male and females aged > 60 years old
* peripheral artery disease at Leriche-Fontaine's stage 2a or 2b
* cognitive functioning to give informed consent identified by a Mini Mental Status Examination score ≥18/30.

Exclusion Criteria:

* peripheral artery disease at Leriche-Fontaine's stage 1
* peripheral artery disease at Leriche-Fontaine's stage 3 or more
* severe cardio-respiratory conditions (e.g. unstable angina; severe heart failure identified by New York Heart Association class III or IV)
* neurological or musculoskeletal conditions (e.g. above knee amputation) contraindicating or inhibiting exercise training.
* very good exercise capacity determined by a 6-minute walking distance > 500 meters.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
6-Minute Walking Test (mobility) | Change at 6-month (end of training) respect to baseline
  Subjects will be instructed to walk as far as possible on a 21m walkway in 6 minutes, with their habitual walking device, with the possibility to slow down and rest if necessary. The total distance walked, the pain-free walking distance, and the perceived exertion at the end of the test will be recorded.

SECONDARY OUTCOMES:
Ankle Brachial Index (hemodynamics) | Change at 6-month (end of training) respect to baseline
  The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). The ABI is calculated by dividing the systolic blood pressure measured at the ankle for both limbs with the patient in supine position by the systolic blood pressure in the arm.
Vascu-QoL-6 (health-related quality of life) | Change at 6-month (end of training) respect to baseline
  This questionnaire consists of 6 items with a score ranging from 1 to 4 examining various aspects of disease-related quality of life. Higher scores correspond to better quality of life.
5-time sit-to-stand test (lower limbs strength) | Change at 6-month (end of training) respect to baseline
  This test consists in moving from a sitting position to a standing position on a 42- cm high chair as quick as possible, for five times, with arms folded across the chest. Time will be taken when the test starts, and when the patient lay his/her buttocks on the chair for the fifth time.
Foot temperature | Change at 6-month (end of training) respect to baseline
  Foot temperature will be noninvasively measured through an infrared thermal imaging camera at the dorsum of each foot at three points
Number and rate of hospitalizations | 6-month, 12-month and 24-month (follow up)
  Number and rate of all-cause hospitalizations within participants will be collected.
Number and rate of mortality | 6-month, 12-month and 24-month (follow up)
  Number and rate of all-cause mortality within participants will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Manfredini, MD, PhD, Principal Investigator — University of Ferrara and University Hospital of Ferrara
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published at the end of the trial after deidentification.
Time Frame: Individual participant data will be available beginning 6 months following study results publication.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Manfredini F, Malagoni AM, Mascoli F, Mandini S, Taddia MC, Basaglia N, Manfredini R, Conconi F, Zamboni P. Training rather than walking: the test in -train out program for home-based rehabilitation in peripheral arteriopathy. Circ J. 2008 Jun;72(6):946-52. doi: 10.1253/circj.72.946. PMID 18503221
- [Background] Treat-Jacobson D, McDermott MM, Bronas UG, Campia U, Collins TC, Criqui MH, Gardner AW, Hiatt WR, Regensteiner JG, Rich K; American Heart Association Council on Peripheral Vascular Disease; Council on Quality of Care and Outcomes Research; and Council on Cardiovascular and Stroke Nursing. Optimal Exercise Programs for Patients With Peripheral Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Jan 22;139(4):e10-e33. doi: 10.1161/CIR.0000000000000623. No abstract available. PMID 30586765
- [Derived] Manfredini F, Lamberti N, Traina L, Zenunaj G, Medini C, Piva G, Straudi S, Manfredini R, Gasbarro V. Effectiveness of Home-Based Pain-Free Exercise versus Walking Advice in Patients with Peripheral Artery Disease: A Randomized Controlled Trial. Methods Protoc. 2021 May 10;4(2):29. doi: 10.3390/mps4020029. PMID 34068534